CLINICAL TRIAL: NCT02103322
Title: A Randomized, Open Label, Two-Treatment, Multiple Dose, Steady State, Two-period, Cross-over, Multi-Centre Comparative Bioequivalence Study of Imatinib Mesylate Tablet 400 mg of Amneal Pharmaceuticals, USA With GLEEVEC® (Imatinib Mesylate) Tablets 400 mg Distributed by Novartis Pharmaceuticals Corporation, East Hanover, New Jersey 07936 in Adult Patients Suffering From Chronic Myeloid Leukemia & Gastrointestinal Stromal Tumor Under Fed Conditions
Brief Title: Comparative Bioequivalence Study in Adult Patients Suffering From Chronic Myeloid Leukemia & Gastrointestinal Stromal Tumor Under Fed Conditions
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Collaborators: Accutest Research Laboratories (I) Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARL/CT/13/001
Record Dates: First submitted 2014-04-01; First posted 2014-04-03 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Myeloid Leukemia; Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imatinib Mesylate Tablets, 400 mg (Experimental): Imatinib Mesylate Tablets, 400 mg. Once daily for 14 days.
  Interventions: Drug: Imatinib Mesylate Tablets, 400 mg
- Gleevec Tablets, 400 mg (Active Comparator): Imatinib Mesylate Tablets, 400 mg. Once daily for 14 days.
  Interventions: Drug: Imatinib Mesylate Tablets, 400 mg

INTERVENTIONS:
Drug: Imatinib Mesylate Tablets, 400 mg — Brown, oval, scored, film coated, beveled edge tablet. Debossed with AN on scored side and 795 on the other side.
  Arms: Imatinib Mesylate Tablets, 400 mg
Drug: Imatinib Mesylate Tablets, 400 mg — Very dark yellow to brownish orange, film-coated tablets, ovaloid, biconvex with bevelled edges, debossed with "400" on one side with score on the other side, and "SL" on each side of the score.
  Other Names: Gleevec
  Arms: Gleevec Tablets, 400 mg

SUMMARY:
To characterize pharmacokinetic profile of test product compared to that of the corresponding reference product in adult patients, who are diagnosed to have Chronic Myeloid Leukemia & Gastrointestinal Stromal Tumor under Fed Conditions.

DETAILED DESCRIPTION:
To characterize pharmacokinetic profile of Imatinib Mesylate tablets EQ 400 mg base of Amneal Pharmaceuticals LLC, compared to that of the reference product - GLEEVEC® (imatinib mesylate) tablets 400 mg in adult patients, who are diagnosed to have CML or GIST and are presently receiving stable dose of imatinib mesylate tablets 400 mg, and assess their bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years (both inclusive) and either sex
* Diagnosed case of Philadelphia chromosome positive (Ph+) CML patients in chronic phase or GIST and presently being treated with imatinib 400 mg tablets.
* Willing to give written informed consent for participation in the study as well as willing and able to comply with study visit schedule and other protocol requirements.
* Female patients of child bearing potential (except for those who have completed one year since menopause or have gone through hysterectomy or bilateral tubal ligation) must have negative serum pregnancy test at the screening, negative urine pregnancy test on check in to housing, must be non-lactating at screening and must agree to use effective contraception (barrier or hormonal) for the study period.

Exclusion Criteria:

* History of hypersensitivity to imatinib mesylate or to any of the excipients as judged by investigator.
* Patient of CML receiving treatment in Myeloid Blast Crisis or Accelerated Phase
* Abnormal laboratory results as below:
* History of a heart failure, renal insufficiency, hypereosinophilic syndrome (HES), myelodysplastic syndrome (MDS)/ myeloproliferative disease (MPD) or acute systemic mastocytosis (ASM).
* History of therapy with any of the following as per timelines before randomization: inducers of CYP3A4 activity and inhibitors of CYP3A4 activity, within 14 days, investigational product/device within last one month
* Alcohol or any drug dependence within past one year.
* Blood donation/loss exceeding 200 ml within last 60 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cmax | Days 5, 6, 7, 12, 13, 14 and 15
  Peak maximum concentration over dosing interval in the steady state
AUC0-tau | Days 5, 6, 7, 12, 13, 14 and 15
  The area under the blood concentration curve versus time, calculated by the trapezoid method, from zero time to the dose interval (tau) in the steady state

SECONDARY OUTCOMES:
Tmax | Days 5, 6, 7, 12, 13, 14 and 15
  The time to reach such peak over dosing interval in the steady state
Cmin | Days 5, 6, 7, 12, 13, 14 and 15
  Minimum concentration established at each dose interval end of the steady state
Cavg | Days 5, 6, 7, 12, 13, 14 and 15
  Average concentration in the steady state (= AUC0-tau / tau)
Swing | Days 5, 6, 7, 12, 13, 14 and 15
  Swing in steady state pharmacokinetics, calculated as (CmaxSS-CminSS)/ CminSS
Fluctuation Rate | Days 5, 6, 7, 12, 13, 14 and 15
  Degree of fluctuation in the steady state pharmacokinetics, calculated as (Cmax-Cmin)/CavSS

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Jani, MD, Principal Investigator — Accutest Research Laboratories (I) Pvt. Ltd.
Locations (5):
- India (5):
  - Kailash Cancer Hospital & Research Centre, Vadodara, Gujurat
  - Srinivasam Cancer Care Hospitals India Pvt., Bangalore, Karnataka
  - Karnataka Caner Hospital, Bengaluru, Karnataka
  - Lokmaya Hospital, Pune, Maharashtra
  - Dr. G Viswanathan Speciality Hospitals, Tiruchirappalli, Tamil Nadu